CLINICAL TRIAL: NCT07156071
Title: 12-Week Serum Efficacy Study
Brief Title: 12-Week Study on the Efficacy of Two Serums in Improving Skin Aging and Tone
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ChinaNorm (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C23005059
Record Dates: First submitted 2025-08-20; First posted 2025-09-04 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Facial Skin Aging and Dullness

STUDY DESIGN:
Intervention Model Description: Participants were assigned in parallel to one of two serum groups (Serum 1 or Serum 2), based on stratification by aging type (early aging or mature aging). The products were applied twice daily over 12 weeks.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Serum 1 Group (Experimental): Participants in this arm applied Serum 1 (Fla#897183 329) to the full face twice daily for 12 weeks. The group included both early aging (18-29 years) and mature aging (30-45 years) subgroups.
  Interventions: Other: Serum 1
- Serum 2 Group (Experimental): Participants in this arm applied Serum 2 (Fla#b50198) to the full face twice daily for 12 weeks. The group included both early aging (18-29 years) and mature aging (30-45 years) subgroups.
  Interventions: Other: Serum 2

INTERVENTIONS:
Other: Serum 1 — Applied topically on the full face in the morning and evening for 12 weeks during the treatment period. Used by participants in the Serum 1 group.
  Arms: Serum 1 Group
Other: Serum 2 — Applied topically on the full face in the morning and evening for 12 weeks during the treatment period. Used by participants in the Serum 2 group.
  Arms: Serum 2 Group

SUMMARY:
This study aims to evaluate the anti-aging and skin tone improvement effects of two facial serums over a 12-week period. It was conducted at a single research center with a 2-week washout period followed by full-face application of the test products for 12 weeks.

A total of at least 120 healthy Chinese female participants aged 18 to 45 were enrolled and divided into two treatment groups:Each group included both early aging (18-29 years) and mature aging (30-45 years) subgroups, with at least 30 participants in each subgroup.

ELIGIBILITY:
Inclusion Criteria:

1. Chinese female aged 18-45 years (evenly split among Early aging [18-29 years] and Mature aging [30-45 years]).
2. All skin types (dry, normal, oily, or mixed).
3. Currently experiencing lack of radiance, roughness, dullness, and fine lines or wrinkles on facial skin as self-claimed.
4. Early aging group (18-29 years): Must present with corresponding severity for the attributes evaluated by Dermatologist, including:

   * Skin smoothness, radiance, dullness: grade between 2 and 6 (scale 0-9);
   * Size of acne marks (PIH): size ≥ 2;
   * Small folds on nasolabial zone: grade between 1 and 3 (Skin Aging Atlas, 0-6 scale, Page 56-57).
5. Mature aging group (30-45 years): Must present with corresponding severity for the attributes evaluated by Dermatologist, including:

   * Skin smoothness, radiance, dullness: grade between 4 and 6 (scale 0-9);
   * Small folds on nasolabial zone: grade between 1 and 4 (Skin Aging Atlas, 0-6 scale, Page 56-57);
   * Forehead wrinkles: grade ≥ 2 (Skin Aging Atlas, 0-8 scale, Page 32-33);
   * Crow's feet wrinkles: grade ≥ 2 (Skin Aging Atlas, 0-6 scale, Page 40-41).
6. Regular user of serum and sunscreen products.
7. Did not participate in any clinical test or cosmetic product test on skin within the last 3 months.
8. No exclusion by dermatologist due to other medical or dermatological reasons.
9. In general good health at the time of the study.
10. Willing and able to participate as evidenced by signing of informed consent and photo release form.
11. Must be willing to comply with all study protocol requirements (including using only the skincare products provided during the study and not taking topical or oral treatments such as retinol, hormones, or antioxidant health supplements).

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2023-11-18 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-03-22 (Actual)

PRIMARY OUTCOMES:
Change in Dermatologist-Assessed Wrinkle Attributes | from Baseline to Week 12
  Crow's feet wrinkles, forehead wrinkles, global wrinkles, small folds on nasolabial zone and global fine lines will be evaluated by dermatologist.
Self-assessment Questionnaire | 12 weeks
  Participants will complete a 5-point self-assessment questionnaire at Timm, T4w, T8w, and T12w, evaluating their perception of skin softness, smoothness, plumpness, elasticity, hydration, oil control, and visible aging signs. Ratings from 4 to 5 will be used to calculate "Top 2 box" percentage.
Change in Dermatologist-Assessed Skin Texture and Quality Attributes | from Baseline to Week 12
  Skin smoothness (visual), skin elasticity, skin softness, skin firmness, skin plumpness, cheek pores will be evaluated by dermatologist.
Change in Dermatologist-Assessed Skin Tone Attributes | from Baseline to Week 12
  Skin radiance, skin translucency, skin pigmentation, skin fairness, skin tone evenness and skin dullness will be evaluated by dermatologist.

SECONDARY OUTCOMES:
Change in Skin Hydration Measured by Corneometer | 12 weeks
Change in Skin Elasticity Measured by Cutometer | 12 weeks
Change in Transepidermal Water Loss (TEWL) Measured by Vapometer | 12 weeks
Change in Facial Image-Based Skin Parameters Using VISIA-CR | 12 weeks
Change in Cheek Skin Surface Condition Using VisioScan VC20 | 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai China-norm Quality Technical Service Co., Ltd., Shanghai, Shanghai 200072, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided